CLINICAL TRIAL: NCT01024348
Title: Open-label Study of the Safety and Effectiveness of Short-term Therapy With Extended-release Tramadol (TRAMADEX-OD) in the Management of Pain After Knee Arthroscopy.
Brief Title: Safety and Effectiveness of Tramadex-OD After Knee Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Yaacov Gozal, MD, Shaare Zedek Medical Center, Jerusalem, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: gozal123456
Record Dates: First submitted 2009-10-13; First posted 2009-12-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Postoperative Pain
Keywords: Surgery, knee arthroscopy; Pain, postoperative; tramadol, extended release
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol; Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tramadex-OD (Active Comparator): Patients will undergo knee arthroscopy under spinal anesthesia without any opioid. 30 minutes prior to surgery and 24 hours afterwards, patients will take a tablet of 100 mg Tramadex-OD. Breakthrough pain will be managed with 1 gr paracetamol (per os) as needed.
  Interventions: Drug: extended-release tramadol
- Control group (Active Comparator): Patients will undergo knee arthroscopy under spinal anesthesia without any opioid.Postoperative pain will be managed throughout the study with 1 gr paracetamol (per os) every 6 hours as required.
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: extended-release tramadol — 30 minutes prior vto surgery and 24 hours afterwards, patients will take a tablet of 100 mg TRAMADEX-OD
  Other Names: Tramadol; Tramal
  Arms: Tramadex-OD
Drug: paracetamol — in the control group, postoperative pain will managed with 1 gr paracetamol (per os) as needed (up to 4 times a day)
  Other Names: Acamol; Acetominophen
  Arms: Control group

SUMMARY:
Extended-release tramadol is indicated for the management of moderate to severe pain in adults who require around-the-clock treatment. It provides an extended duration of action, more constant plasma concentrations, a reduced dosing frequency, and the potential for improved compliance and therapeutic outcomes.

The present study was designed to evaluate the safety and effectiveness of this medication in the treatment of early postoperative pain after knee arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Men and nonpregnant women
* Age: 18-65 years
* ASA classification I or II
* ambulatory knee arthroscopy under spinal anesthesia

Exclusion Criteria:

* Pregnancy
* Intolerance to any opioid, tramadol or paracetamol
* spine surgery in the past
* renal or hepatic impairment
* cardiac or respiratory conditions that put the patient at risk for respiratory depression
* patients receiving: monoamine oxidase inhibitors, carbamazepine, quinidine, selective serotonin reuptake inhibitors or tricyclic antidepressants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Safety and effectiveness of TRAMADEX-OD will be evaluated by recording adverse events and using a visual analogue score for pain evaluation | up to 48 hours

SECONDARY OUTCOMES:
Patient satisfaction will be evaluated by a telephone interview | up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yaacov Gozal, MD, Principal Investigator — Shaare Zedek Medical center, Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel